CLINICAL TRIAL: NCT05593861
Title: Assessment of Enhanced Recovery After Surgery Implementation at Pediatric Surgery Practices in Mainland China: Based on a Survey of Performing Congenital Biliary Dilatation Operations
Brief Title: Assessment of Enhanced Recovery After Surgery Implementation at Pediatric Surgery Practices in Mainland China
Status: Completed | Type: Observational
Sponsor: Weibing Tang (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Doctor, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Other Study IDs: NanjingCH13170
Record Dates: First submitted 2022-07-25; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: ERAS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This investigation was conducted on chief surgeons at each center.: This investigation was conducted on chief surgeons at each center.

SUMMARY:
Enhanced recovery after surgery (ERAS) is a new mode to optimize perioperative management, the core of which is to reduce perioperative physiological and psychological trauma and stress damage, and accelerate postoperative rehabilitation. ERAS has been gradually introduced in pediatric surgery in recent years, however, there are limited reports on its overall implementation. We aimed to determine the popularity of ERAS among pediatric populations in mainland China.

DETAILED DESCRIPTION:
The application of ERAS in children with congenital biliary dilatation (CBD) was investigated. A total of 31 province-level administrative regions in mainland China were involved and each of them had at least one participating center. A questionnaire was designed to assess the baseline adherence of 17 recovery elements and chief pediatric surgeons at each center were invited to complete.

ELIGIBILITY:
Inclusion Criteria:

* chief pediatric surgeons at each center

Exclusion Criteria:

* Incomplete questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chief pediatric surgeons at each center
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Element adherence | immediately after all the questionnaires are collected
  Adherence to an element was determined if the frequency of practice reached specific thresholds as defined.

SECONDARY OUTCOMES:
Factors associated with baseline ERAS utilization | immediately after all the questionnaires are collected
  Factors associated with baseline ERAS utilization

OTHER OUTCOMES:
Barriers to implementation | immediately after all the questionnaires are collected
  Barriers to implementation
Outcomes of concern | immediately after all the questionnaires are collected
  Outcomes of concern

CONTACTS AND LOCATIONS:
Overall Officials: Hua Xie, M.M., Principal Investigator — Department of pediatric Surgery, Children's Hospital of Nanjing Medical University, Nanjing, China.
Locations (1):
- NJMU, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Vacek J, Davis T, Many BT, Close S, Blake S, Hu YY, Holl JL, Johnson J, Strople J, Raval MV. A baseline assessment of enhanced recovery protocol implementation at pediatric surgery practices performing inflammatory bowel disease operations. J Pediatr Surg. 2020 Oct;55(10):1996-2006. doi: 10.1016/j.jpedsurg.2020.06.021. Epub 2020 Jun 27. PMID 32713714